CLINICAL TRIAL: NCT00440843
Title: Efficacy of Olanzapine in Improving Task Engagement in Schizophrenia
Brief Title: Zyprexa and Task Engagement in Schizophrenia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: Clinical Trials Network of Columbia U, Cornell U, and NY Presbyterian Hospital (Network); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jimmy Choi, Assistant Professor, VA Connecticut Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JC0002; F1D-US-X282
Record Dates: First submitted 2007-02-25; First posted 2007-02-27 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; attention; task engagement; antipsychotics; cognition; cognitive rehabilitation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OLZ (Experimental)
  Interventions: Drug: Olanzapine (Zyprexa)
- Typicals (Active Comparator)
  Interventions: Drug: Typicals

INTERVENTIONS:
Drug: Olanzapine (Zyprexa) — OLZ
  Arms: OLZ
Drug: Typicals — Stay on typicals regimen
  Arms: Typicals

SUMMARY:
Individuals with schizophrenia frequently have impairments in attention. These impairments have been shown to be related to overall functioning. Some research suggests that Olanzapine may be associated with improvement in various aspects of attention. The primary purpose of this study is to determine whether switching from a typical antipsychotic to Olanzapine improves task engagement. Individuals who taking typical antipsychotics will be randomly assigned to either 1) remain on their typical antipsychotic medications, or 2) be switched from their typical antipsychotic medications to Olanzapine. All participants will be enrolled in a twice-weekly 20 session cognitive training program that is specifically designed to target attention deficits and promote active engagement. Improvements in attention will be compared between individuals who remained on their typical antipsychotic medications and those that were switched to Olanzapine.

DETAILED DESCRIPTION:
Objectives: Olanzapine (OLZ) has emerged as one of the promising pharmacologic interventions that not only improves psychotic symptoms but may also target ability to sustain attention on cognitive tests. Pupillary response, as measured by degree of pupil constriction, and visual scanning patterns are unique methods of quantifying attention by gauging the level of psychophysiologic engagement on a visual task. It is reasonable to expect that if a treatment for attention problems is effective, then this will be reflected in more efficient allocation of psychophysiologic attentional resources as measured by pupillometry. Primary purpose of this pilot study is to demonstrate efficacy of switching to OLZ for improving task engagement in schizophrenia. Secondary objectives are to demonstrate improved attention in response to OLZ translates to improved attentional allocation strategies and vocational readiness, and demonstrate efficacy of OLZ as agent that enhances ability to benefit from cognitive training. The proposed study will examine functional implications of improved attention in patients taking OLZ, and it will test the hypothesis that mechanism of this functional improvement is through process of engagement as measured by pupillometry and functional behavioral measures.

Research Design and Methodology: This is an industry-sponsored, investigator initiated trial with 18 patients in an open-label design over 24-month period. Participants will be adult outpatients (ages 18 to 55) with a diagnosis of schizophrenia or schizoaffective disorder who are on any regimen of "typical" antipsychotics. They will be randomly assigned to one of two conditions: 1) Olanzapine Group (OLZ-G). Subjects assigned to the OLZ condition will be switched to OLZ from their previous medication so OLZ is the only antipsychotic medication part of their regimen. Following switch to OLZ, subjects will be enrolled in a twice weekly, 20-session cognitive training program that is specifically designed to target attention deficits and promote active engagement. 2) "Typicals" Group (TYP-G). Subjects assigned to the "typicals" condition will continue with their medication regimen throughout the course of the study as they are enrolled in the same cognitive training program. Research questions are: Compared to participants on any combination of "typical" medications, we hypothesize that persons with schizophrenia on OLZ will (a) show significantly improved performance on psychophysiologic measure of task engagement, (b) show greater engagement in cognitive training, and (c) show greater improvement in attention on vocational task. Primary efficacy measure will be an ASL H6 Series head-mounted optics pupillometer to measure task engagement as function of pupil dilation and visual scanning patterns. Secondary efficacy measures will include computer software specifically developed to assess on-task behavior on computer exercises, brief neuropsychological test battery, global behavior and symptom inventories, and functional assessment of treatment motivation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Current medication regimen that includes any combination of first generation neuroleptics, for at least 30 days
* Referring psychiatrist agrees to transfer primary psychiatric care and medication prescription to the study doctor, for the duration of patient's participation in the study

Exclusion Criteria:

* Significant auditory/visual impairment that would interfere with study procedures
* Lack of aptitude in English that may interfere with the administration of the tests
* Current use of psychoactive substances that may affect attention (e.g. Amoxetine, Methylphenidate)
* Deviations from the prescription regimen not approved by study doctor
* Changes in the regimen of antipsychotics not included in the study's protocol
* Chart diagnosis of any other medical or neuropsychiatric illnesses known to impair brain function (e.g. mental retardation, traumatic brain injury, seizure disorder).
* Pregnant or breast-feeding females.
* Use of alcohol or drugs 4 weeks prior to beginning of study.
* For participants with history of substance dependence (excluding nicotine and caffeine) use of illicit substances (e.g. marijuana or crack) during study participation.
* Use of a depot antipsychotic within 4 weeks prior to baseline
* History or evidence of a medical or neurological condition that would expose the subject to an undue risk of a significant adverse event or interfere with study assessments
* Clinically significant abnormal laboratory test results at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pupillometry | Baseline, post

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Choi, Psy.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States